CLINICAL TRIAL: NCT06589726
Title: A Single-Dose, Randomized, Double-Blind, Placebo- and Positive-Controlled, 4-Way Crossover Study to Evaluate the Effect of Enpatoran on the QTc (Corrected QT) Interval in Healthy Adult Participants
Brief Title: A TQT Study to Investigate the Effect of Enpatoran on Cardiac Repolarization in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS200569_0065; 2024-512841-17-00 (Other: EU CT Number)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Healthy
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence 1: A-B-C-D (Experimental): Participants will receive a single oral dose of placebo matched to enpatoran (Treatment A) in treatment period 1, followed by a single oral dose of moxifloxacin tablet (Treatment B) in treatment period 2, followed by a single oral low dose of enpatoran tablet (Treatment C) in treatment period 3, followed by a single oral high dose of enpatoran tablet (Treatment D) in treatment period 4. There will be a washout period of at least 10 days between each treatment period.
  Interventions: Drug: Placebo; Drug: Moxifloxacin; Drug: Enpatoran low dose; Drug: Enpatoran high dose
- Treatment Sequence 2: B-D-A-C (Experimental): Participants will receive a single oral dose of moxifloxacin tablet (Treatment B) in treatment period 1, followed by a single oral high dose of enpatoran tablet (Treatment D) in treatment period 2, followed by a single oral dose of placebo matched to enpatoran (Treatment A) in treatment period 3, followed by a single oral low dose of enpatoran tablet (Treatment C) in treatment period 4. There will be a washout period of at least 10 days between each treatment period.
  Interventions: Drug: Placebo; Drug: Moxifloxacin; Drug: Enpatoran low dose; Drug: Enpatoran high dose
- Treatment Sequence 3: C-A-D-B (Experimental): Participants will receive a single oral low dose of enpatoran tablet (Treatment C) in treatment period 1, followed by a single oral dose of placebo matched to enpatoran (Treatment A) in treatment period 2, followed by a single oral high dose of enpatoran tablet (Treatment D) in treatment period 3, followed a by single oral of moxifloxacin tablet (Treatment B) in treatment period 4. There will be a washout period of at least 10 days between each treatment period.
  Interventions: Drug: Placebo; Drug: Moxifloxacin; Drug: Enpatoran low dose; Drug: Enpatoran high dose
- Treatment Sequence 4: D-C-B-A (Experimental): Participants will receive a single oral high dose of enpatoran tablet (Treatment D) in treatment period 1, followed by a single oral low dose of enpatoran (Treatment C) in treatment period 2, followed by a single oral dose of moxifloxacin tablet (Treatment B) in treatment period 3, followed by a single oral dose of placebo matched to enpatoran (Treatment A) in treatment period 4. There will be a washout period of at least 10 days between each treatment period.
  Interventions: Drug: Placebo; Drug: Moxifloxacin; Drug: Enpatoran low dose; Drug: Enpatoran high dose

INTERVENTIONS:
Drug: Placebo — Participants will receive a single oral dose of placebo matched to enpatoran in either of treatment period 1, 2, 3 and 4.
Drug: Moxifloxacin — Participants will receive a single oral dose of moxifloxacin tablet (Treatment B) in either of treatment period 1, 2, 3 and 4.
Drug: Enpatoran low dose — Participants will receive a single oral low dose of enpatoran tablet (Treatment C) in either of treatment period 1, 2, 3 and 4.
  Other Names: M5049
Drug: Enpatoran high dose — Participants will receive a single oral high dose of enpatoran tablet (Treatment D) in either of treatment period 1, 2, 3 and 4.
  Other Names: M5049

SUMMARY:
The purpose of this study is to assess potential effects of enpatoran on cardiac repolarization (i.e. prolongation of QT interval).

ELIGIBILITY:
Inclusion criteria:

* Participants are overtly healthy, as determined by medical evaluation, including no clinically significant abnormality identified on medical history, physical examination, vital signs, 12-lead ECG, or laboratory evaluation and no active clinically significant disorder, condition, infection, or disease that would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion
* Participants have a body weight within the range 50.0 to 100.0 kilograms (kg) (inclusive) and body mass index (BMI) within the range 19.0 to 30.0 kilograms per square meter (kg/m^2) (inclusive)
* Other protocol defined inclusion criteria could apply

Exclusion criteria:

* History or presence of clinically relevant respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, musculoskeletal, genitourinary, immunological, dermatological, connective tissue, psychiatric (due to rare risk of hallucinations, agitation, and activation of psychosis), and other diseases or disorders, and epilepsy, as determined by medical evaluation
* Individuals with diagnosis of hemochromatosis, Wilson´s disease, alpha 1 antitrypsin deficiency, or any other chronic liver disease including Gilbert's disease
* Prior history of cholecystectomy or splenectomy, and any clinically relevant surgery within 6 months prior to the first administration of study intervention
* History of malignancy (e.g. hematologic, skin, solid tumor) less than or equal to (<=) 10 years prior to Screening
* History of chronic or recurrent acute infection or any bacterial, viral, parasitic, or fungal infections within 30 days prior to Screening and at any time between Screening and admission to CRU, or hospitalization due to infection within 6 months prior to the first administration of study intervention
* History of shingles within 12 months prior to Screening
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Placebo-Corrected Change from Baseline in Heart Rate-Corrected QT Interval by Fridericia's Formula (QTcF) for Enpatoran | Pre-dose on Day 1 (baseline) up to 24 hours post-dose

SECONDARY OUTCOMES:
Placebo-Corrected Change from Baseline in Heart Rate-Corrected QT Interval by Fridericia's Formula (QTcF) for Moxifloxacin | Pre-dose on Day 1 (baseline) up to 24 hours post-dose
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to approximately 72 days
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) by Severity | Up to approximately 72 days
Number of Participants with Abnormal Laboratory Parameters, Vital Signs and 12-Lead Electrocardiogram (ECG) Findings | Up to approximately 72 days
ECG Parameters: QT Interval, heart rate-corrected QT interval (QTc), individual corrected QT interval (QTcI), PR Interval, QRS interval and RR Interval | Pre-dose up to 24 hours post-dose
ECG Parameter: Heart Rate (HR) | Pre-dose up to 24 hours post-dose
Number of Participants with T-wave Morphology Changes and U-wave Presence | Pre-dose up to 24 hours post-dose
Pharmacokinetic (PK) Plasma Concentrations of Enpatoran | Pre-dose up to 24 hours post-dose
Pharmacokinetic (PK) Plasma Concentrations of Moxifloxacin | Pre-dose up to 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200569_0065
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html